CLINICAL TRIAL: NCT02317640
Title: Testosterone Replacement Therapy in Combination With Electrical Stimulation and Standing: Effect on Muscle and Bone in Spinal Cord Injured Males.
Brief Title: TRT in Combination With Electrical Stimulation and Standing: Effect on Muscle and Bone in Spinal Cord Injured Males
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gail Forrest, Principal Investigator, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DOD SC130243
Record Dates: First submitted 2014-12-06; First posted 2014-12-16 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Spinal Cord Injury
Keywords: Testosterone; Electrical Stimulation; Stand Training
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Stand Training Alone (Active Comparator): Standing training will be prescribed 3 days/week (1.5 hours/sessions) for 60 sessions. All individuals randomized to stand training will train with BWST with manual assistance and will undergo a stand evaluation. During the evaluation the participants will be placed on the treadmill in an upright position and suspended in a harness by an overhead cable (i.e. BWST). A trainer will be positioned to assist the participant while standing and to provide manual assistance if needed. The amount of BWS and level of assistance given for each body segment will be recorded. The BWS level at which the participant can independently support good standing posture will also be recorded. Standing time while on treadmill and overground will be recorded daily as part of the training sessions.
  Interventions: Other: Stand Training
- ST with placebo or testosterone (Experimental): Stand Training as described above with Placebo or testosterone Gel applied by a pump. After a baseline testing period, TRT will begin in the treatment groups by application of a daily dose of 40.5 mg of testosterone or placebo gel. The gel is to be applied to the upper arms and shoulders and is absorbed and eliminated over the course of a day. To ensure proper dosing serum T concentration will be assessed at screening, baseline, 2 weeks, 1 month and 3 month time points. As such, follow-up with the participant will be necessary to determine the correct replacement dose of TRT, and adjustment of dose if needed, (i.e. 40.5 mg up to 81 mg of gel). If serum T levels are not within normal range at the 2 week time point, the dose will be increased in increments of 20.25 mg up to 81 mg.
  Interventions: Drug: Testosterone Gel applied by a pump; Other: Stand Training
- ST with Placebo or Testosterone and ES (Experimental): Stand Training described above with Placebo or testosterone gel applied by a pump. Electrical stimulation will be applied via bifurcated leads and self-adhesive reusable surface electrodes. The electrodes will be applied over the motor points (both legs) on the following muscles: gluteus maximus (GL), rectus femoris (RF), biceps femoris (BF), gastrocnemei (GC), and anterior tibialis (TA) of both legs. Two electrodes will be used for each muscle. One "RT300 portable stimulator" (Restorative Therapies, Inc., Baltimore, MD) will be used to induce the electrical stimulation with 10 sets of electrodes for stimulation.
  Interventions: Drug: Testosterone Gel applied by a pump; Other: Stand Training; Device: Electrical Stimulation
- ST with ES (Experimental): Stand Training as described above in Stand Training alone and Electrical Stimulation as described above in ST with Placebo or Testosterone and ES.
  Interventions: Other: Stand Training; Device: Electrical Stimulation

INTERVENTIONS:
Drug: Testosterone Gel applied by a pump — After being diagnosed with low testosterone levels the participant will be given a 30-day supply of the Testosterone/placebo gel (40.5 mg/day). The gel is to be applied every morning on clean and dry area of skin of the upper arms and shoulders.
  Other Names: Androgel 1.62%
  Arms: ST with Placebo or Testosterone and ES; ST with placebo or testosterone
Other: Stand Training — Stand training with BWST with manual assistance. Participant is placed on treadmill in an upright position and suspended in a harness by an overhead cable. A trainer will aid the participant in pelvis and trunk stabilization, by applying anterior forces at the pelvis and/or posterior forces at the shoulders and ensure that the trunk and pelvis are not flexed or hyper-extended.
  Other Names: Locomotor Training
Device: Electrical Stimulation — Electrical Stimulation (ES) will be applied via bifurcated leads and self-adhesive reusable surface electrodes. The electrodes will be applied over the motor points of both legs. Two electrodes will be used for contracting each muscle.
  Other Names: ES
  Arms: ST with ES; ST with Placebo or Testosterone and ES

SUMMARY:
The aim of this study is to understand what happens to muscle and bone in spinal cord injured males after four months of training using stand training, with body weight support (BWS), with testosterone replacement therapy (TRT), and electrical stimulation (ES). Specifically, researchers will investigate nerve, muscle, and bone changes in the lower limbs in response to stand training and ES when combined with TRT compared to i) standing alone with TRT; ii) stand training alone with placebo; iii) stand training alone and ES with placebo.

DETAILED DESCRIPTION:
Primary Aim:

To assess the effects of our novel tri combination Activity-Dependent Rehabilitation model approach on muscle volume of the lower limbs.

Secondary Aims:

i) To better define the mechanisms that contribute to changes in muscle.

Preliminary data from animal studies have shown increased expression of Activin receptor IIB and increased nuclear localization of Smad2 and Smad3 after SCI and that these adverse changes are reversed by androgens. Additional studies will examine mRNA levels for myostatin, its receptor and its inhibitors (e.g., follistatins) and determine nuclear levels of Smad2 and Smad3. We will also measure resting energy expenditure to confirm that changes in muscles mass correspond to anticipated metabolic effects.

ii) To evaluate the changes in bone and bone structure with Stand Training with TRT and ES.

Individuals with SCI not only lose motor and/or sensory function, they experience dramatic muscle and bone loss. Locomotor training, an activity-based intervention that engages the neuromuscular system below the level of lesion for standing and walking enhances EMG activity and has shown modest improvements in muscle without any attenuation in bone density [172-177]. Dynamic stand training, an important component of locomotor training, provides sensory feedback related to standing and bilateral weight bearing, resulting in bilateral muscle activation via central pathways through the spinal cord [161,178-181]. Thus, the stand retraining component provides a physiologically relevant multi-muscle activation through central pathways, dynamic gravity opposed loading of the legs and additional task specific activation of the muscles [161,162,179]. Functional electrical stimulation is a method of exercise that has been employed in the SCI population and has demonstrated success in improving muscle, with less conclusive evidence for its effect on bone albeit there has been speculation that although slowing or preventing bone loss may be feasible after SCI, reversing such bone loss (i.e. restoring bone) is not possible, although the evidence is primarily from applying FES to single muscles [151,171]. TRT has been shown to offer a logical, efficacious, and cost-effective intervention to, in part, counteract these untoward body composition, metabolic, and functional sequelae of relative hypogonadism in those with chronic SCI [37]. In addition, testosterone alone has been shown to increase muscle mass, muscle strength, and bone in androgen-deficient men and older men with low testosterone levels [182,183]. The model of compressive loads generated during the combination of stand retraining and multi muscle ES will be multi-directional and will increase muscle strength and the forces applied to the hip, femur and tibia bones. We anticipate that the model of standing plus TRT will increase muscle mass and strength more than standing alone. The combination of multi muscle TRT+ES while stand training will further increase muscle strength compared to either arm alone, resulting in an increased synergistic response of benefit which will surpass the threshold needed to significantly increase bone restoration [102,184,185].This novel tri-combination synergistic approach of TRT, ES, and Stand Training is being hypothesized to increase muscle mass and strength to a greater extent than that of each alone or than that of only two of these interventions. Measurements of muscle torques will be obtained to demonstrate a quantifiable relationship between muscle strength and bone mass.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a male between 18 and 58 years old;
2. Must have a spinal cord injury at a neurological level of injury between the C6-T10 level and an impairment grade A, B, or C, according to the American Spinal Injury Association (ASIA) Impairment Scale. If a person with quadriplegia their motor level will be used instead of neurological level. As a quadraplegic the motor level must be between C6-T10;
3. Must be able to tolerate electrical stimulation and must show visible muscle contraction to an electrical stimulus;
4. Must be wheelchair reliant for more than 75% of the time;
5. Must have low testosterone levels (300-325 ng/dL) as determined by a blood test done at the baseline study visit.

Exclusion Criteria:

1. Taking spasticity medication (i.e., baclofen). It may be possible that participant can be weaned off of the spasticity medication prior to starting entry into the study. This would be under the guidance of the study physician.
2. Less than 6 months or greater than 10 years post injury;
3. A score >3 on the Modified Ashworth Scale as determined by study staff;
4. Bone density measurement for the knee is at or below .5755 gm/cm2 as recorded by study staff;
5. Weigh more than 225 lbs;
6. Taller than 6 feet 3 inches;
7. Presence of a cardiovascular disease;
8. Presence of pulmonary disease;
9. Presence of recent lower limb fractures;
10. Presence of severe contractures;
11. Presence of lower extremity deep vein thrombosis (within the last three months) or other major medical illness;
12. Taking medications known to influence bone metabolism as determined by study staff review of medications;
13. A major gastrointestinal problem such as swallowing or gastrointestinal reflux disease;
14. Heart rate or rhythm problems;
15. A pacemaker;
16. Had spinal fusion, must have approval from the referring physician to receive ES - assisted standing prior to acceptance into the study;
17. As determined by study staff and review of medications, taking medication known to affect my level of testosterone;
18. A PSA greater than or equal to 4.0 ng/ml as determined by blood tests during screening visit;
19. An elevated PSA or asymmetry or hardening of prostate as determined by blood tests and digital rectal examination at screening visit.
20. Any known heart or blood vessel problems (cardiovascular disease)
21. An acute illness of any cause;
22. History of anabolic steroid use as determined by study staff review of participant's medical records;
23. Have a hematocrit greater than or equal to 55 as measured by the study team.
24. Have an abnormal liver function test from the hepatic panel (greater than 2.5 times the normal value) as measured by the study team;
25. Have an abnormal digital rectal exam (DRE) at baseline suggestive of malignancy;
26. Currently abuse alcohol or drugs;
27. Have a significant psychological disorder;
28. Have a history of or a current malignancy;
29. Wish to contribute to the conception of a child.

If any of the following occurs in the experimental group following initiation of testosterone replacement therapy participation will be terminated.

1. Hematocrit greater than or equal to 55;
2. Abnormal liver function test from the hepatic panel (greater than 2.5 times the normal value);
3. Worsening of any sleep disorder, as determined by the Investigators;
4. A PSA greater than or equal to 4.0 ng/ml;
5. Worsening of mood disorders; i.e. anger and depression as determined by the investigators;
6. Planning to contribute to the conception of a child during the study period.
7. Have participated in an electrical stimulation or TRT study in the previous 3 months.

Ages: 18 Years to 58 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Muscle Volume (percent change in muscle volume for the bilateral thigh) | 38 weeks
  Muscle volume will be measured in the thigh. The percent change in muscle volume for the bilateral thigh will be compared to before the intervention to after the intervention.

SECONDARY OUTCOMES:
Change in Muscle (increase in muscle torque) | 38 weeks
  To assess whether the tri-combination of stand training with TRT and ES will lead to increased muscle strength and contractile elements of muscle as shown by an increase in muscle torque.
Change in Bone (BMD of the proximal tibia and distal femur) | 38 Weeks
  To evaluate change in bone and bone structure with stand training with TRT and ES will include BMD of the proximal tibia and distal femur; these are the most common sites for fracture and may also respond faster to intervention. Other secondary outcome measures will be BMD at the hip, cortical and trabecular bone with 3-D volumetric measurements, and bone markers for formation and resorption.

CONTACTS AND LOCATIONS:
Overall Officials: Gail F Forrest, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States